CLINICAL TRIAL: NCT02282657
Title: Pilot Feasibility and Safety Study on Low-flow Extracorporeal CO2 Removal in Patients With Moderate ARDS to Enhance Lung Protective Ventilation
Brief Title: Strategy of UltraProtective Lung Ventilation With Extracorporeal CO2 Removal for New-Onset Moderate to seVere ARDS
Acronym: SUPERNOVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPERNOVA
Record Dates: First submitted 2014-10-21; First posted 2014-11-04 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Moderate Acute Respiratory Distress Syndrome
Keywords: extracorporreal; CO2 removal; ARDS; lung; Protective ventilation
MeSH Terms: interventions — Neuromuscular Blocking Agents; Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One single arm (Experimental): Procedure: Baseline ventilator settings will be established per the EXPRESS protocol: VT = 6 mL/kg (ideal body weight); inspiratory flow will be set at 50-70 L/min resulting in an end-inspiratory pause of 0.2-0.5 sec, I:E ratio 1:1 to 1:3, PEEP set so that the plateau pressure (Pplat), measured during the end-inspiratory pause of 0.2 to 0.5 s, will be within the following limits: 28 cm H2O ≤ Pplat ≤ 30 cm H2O; Set RR to 20-35 to maintain approximately the same minute ventilation as before study initiation. Baseline ventilator settings will be maintained for a 2-hour run-in time (time to setup ECCO2R devices). Use heated humidifiers for gas humidification and minimize instrumental dead space. ECCO2R will be initiated during the 2-hour run-in time. Neuromuscular blocking agents (NMBA) will be used. EtCO2 will be monitored. RR will be kept what it was at Baseline. Sweep gas flow will be adapted. Ventilation will be adapted. Respiratory rate will be adapted.
  Interventions: Device: ECCO2R will be initiated during the 2-hour run-in time; Other: Neuromuscular blocking agents (NMBA); Device: Ventilation; Other: Level of carbon dioxide released at the end of expiration; Other: Respiratory Rate; Other: Sweep gas flow; Other: Ventilation will be adapted; Other: Respiratory rate will be adapted

INTERVENTIONS:
Device: ECCO2R will be initiated during the 2-hour run-in time — A single (15.5 to 19 Fr) veno-venous ECCO2R catheter will be inserted percutaneously (jugular vein strongly suggested).
  Catheters should be rinsed with heparinized saline solution before insertion Once the catheter has been inserted each line will be filled with an heparinized saline solution before its connection to the extracorporeal circuit The ECCO2R circuit will be connected to the catheter and blood flow set, depending on the device, up to 1000 mL/min.
  Initially, sweep gas flow through the ECCO2R device will be set at zero (0 LPM) such as to not initiate CO2 removal through the device.
  Anticoagulation will be maintained with unfractionated heparin to a target aPTT of 1.5 - 2.0X baseline. A bolus of heparin is suggested at the time of cannulation.
Other: Neuromuscular blocking agents (NMBA) — Patients will receive NMBA starting in the run-in period and continued for the first 24 hours and thereafter will be directed by the attending physician
Device: Ventilation — Following the 2-hour run-in time, VT will be reduced gradually to 5 mL/kg. Sweep gas initiated then VT decreased to 4.5 then 4 mL/kg and PEEP adjusted to reach 23 ≤ Pplat ≤ 25 cm H2O.
Other: Level of carbon dioxide released at the end of expiration — EtCO2 will be monitored for safety purposes. Blood gases will be analyzed 20-30 minutes after each VT reduction
Other: Respiratory Rate — RR will be kept what it was at baseline
Other: Sweep gas flow — Sweep gas flow will be adapted to maintain the same EtCO2
Other: Ventilation will be adapted — If PaCO2> 75 mmHg and/or pH < 7.2, despite respiratory rate of 35/min and optimized ECCO2R, VT will be increased to the last previously tolerated VT.
Other: Respiratory rate will be adapted — If PaCO2 remains within the target range, respiratory rate will be progressively decreased to a minimum of 15/ min and facilitated by increases in sweep flow.

SUMMARY:
Pathophysiological, experimental and clinical data suggest that an '"ultraprotective" mechanical ventilation strategy may further reduce VILI and ARDS-associated morbidity and mortality. Severe hypercapnia induced by VT reduction in this setting might be efficiently controlled by ECCO2R devices. A proof-of-concept study conducted on a limited number of ARDS cases indicated that ECCO2R allowing VT reduction to 3.5-5 ml/kg to achieve Pplat<25 cm H2O may further reduce VILI.

DETAILED DESCRIPTION:
Over the past few decades, highly significant progress has been made in understanding the pathophysiology of the acute respiratory distress syndrome (ARDS). Recognition of ventilation-induced lung injuries (VILI) has led to the radical modification of the ventilatory management of these patients. The landmark trial by the ARDSnet trial group demonstrated in 2000 that ventilating ARDS patients with a low tidal volume (VT) of 6 ml/kg (calculated from predicted body weight), and with a maximum end-inspiratory plateau pressure (Pplat) of 30 cmH2O decreased mortality from 39.8% (in the conventional arm treated with a VT of 12 ml/kg PBW) to 31% . However, recent studies have shown that lung hyperinflation still occurs in approximately 30% of ARDS patients even though they are being ventilated using the ARDSNet strategy. Additionally, Hager and coworkers found that mortality decreased as Pplat declined from high to low levels at all levels of Pplat on the data collected by the "ARDSNet" trial group. Their analysis suggested a beneficial effect of VT reduction even for patients who already had Pplat<30 cm H2O before VT reduction.Similar observation was also recently reported by Needham et al on a cohort of 485 patients with ARDS. Because VT reduction to <6 ml/kg to achieve very low Pplat may induce severe hypercapnia and may cause elevated intracranial pressure, pulmonary hypertension, decreased myocardial contractility, decreased renal blood flow, and the release of endogenous catecholamines, this strategy using "ultraprotective" MV settings is not possible for most patients on conventional mechanical ventilation for moderate to severe ARDS.

Extracorporeal carbon dioxide removal (ECCO2R) may be used in association with mechanical ventilation to permit VT reduction to <6 ml/kg and to achieve very low Pplat (20-25 cm H2O). In an observational study conducted in the 80's, Gattinoni showed that use of venovenous ECCO2R at a flow of 1.5-2.5 l/min in addition to quasi apneic mechanical ventilation with peak inspiratory pressures limited to 35-45 cmH2O and PEEP set at 15-25 cmH2O resulted in lower than expected mortality in an observational cohort of severe ARDS patients. However, a randomized, controlled single-center study using that same technology and conducted in the 1990s by Morris's group in Utah was stopped early for futility after only 40 patients had been enrolled and failed to demonstrate a mortality benefit with this device (58% in the control group vs. 70% in the treatment group).

In recent years, new-generation ECCO2R devices have been developed. They offer lower resistance to blood flow, have small priming volumes and have much more effective gas exchange. With ECCO2R the patient's PaCO2 is principally determined by the rate of fresh gas flow through the membrane lung. In an ECCO2R animal model, CO2 removal averaged 72±1.2 mL/min at blood flows of 450 mL/min, while CO2 production by the lung decreased by 50% with reduction of minute ventilation from 5.6 L/min at baseline to 2.6 L/min after insertion of the device. Lastly, Terragni et al (15)demonstrated that ECCO2R could improve pulmonary protection by allowing very low tidal volume ventilation (3.5-5 ml/kg of PBW) in a proof-of-concept study of ten patients with ARDS. This strategy was also associated with a significant decrease in pulmonary inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation with expected duration of >24h
* Moderate ARDS according to the Berlin definition(16) PaO2/FiO2: 200-100 mmHg, with PEEP ≥ 5 cmH2O

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Decompensated heart insufficiency or acute coronary syndrome
* Severe COPD
* Major respiratory acidosis PaCO2>60 mmHg
* Acute brain injury
* Severe liver insufficiency (Child-Pugh scores >7) or fulminant hepatic failure
* Heparin-induced thrombocytopenia
* Contraindication for systemic anticoagulation
* Patient moribund, decision to limit therapeutic interventions
* Catheter access to femoral vein or jugular vein impossible
* Pneumothorax
* Platelet <50 G/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Achievement of VT reduction to 4 mL/kg while maintaining pH and PaCO2 to ± 20% of baseline values obtained at VT of 6 mL/kg. | maximum 28 days

SECONDARY OUTCOMES:
Assessment of the changes in pH/ PaO2 /PaCO2 | maximum 28 days
  Assessment of the changes in pH/ PaO2 /PaCO2
Device CO2 clearance in the first 24 hours of ECCO2R | maximum 28 days
  device CO2 clearance in the first 24 hours of ECCO2R following VT reduction from 6 mL/kg to 4 ml/kg.
Amount of CO2 removed by the ECCO2R device | maximum 28 days
  During the first 12 hours (every hour) Thereafter at least twice daily at 08:00 ± 2 hours and 20:00 ± 2 hours.
Evaluation of lung recruitment/derecruitment (FRC measurement by the ventilator, ECHO-LUS…) | maximum 28 days
The frequency of serious adverse events (SAE). | maximum 28 days
  Examples of adverse events that are expected in the course of ARDS include transient hypoxemia, agitation, delirium, nosocomial infections, intolerance of gastric feeding, or skin breakdown. Such events, which are often the focus of prevention efforts as part of usual ICU care, will not be considered reportable adverse events unless the event is considered by the investigator to be associated ECCO2-R, or events that are unexpectedly severe or frequent for an individual patient with ALI (Acute Lung Injury).

CONTACTS AND LOCATIONS:
Overall Officials: Alain COMBES, PhD, Principal Investigator — La pitié-Salpétrière Hospital; Marco RANIERI, PhD, Principal Investigator — University of Turin S.Giovanni Battista Molinette Hospital
Locations (1):
- selected ICUs for the pilot phase, Different Locations and Several Countries, Belgium

REFERENCES:
- [Background] Dreyfuss D, Ricard JD, Saumon G, (2003) On the physiologic and clinical relevance of lung-borne cytokines during ventilator-induced lung injury. Am J Respir Crit Care Med 167: 1467-1471. Rouby JJ, Puybasset L, Nieszkowska A, Lu Q, (2003) Acute respiratory distress syndrome: lessons from computed tomography of the whole lung. Crit Care Med 31: S285-295. Dreyfuss D, Saumon G, (1998) Ventilator-induced lung injury: lessons from experimental studies. Am J Respir Crit Care Med 157: 294-323. Frank JA, Parsons PE, Matthay MA, (2006) Pathogenetic significance of biological markers of ventilator-associated lung injury in experimental and clinical studies. Chest 130: 1906-1914. The Acute Respiratory Distress Syndrome Network. (2000) Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med 342: 1301-1308. Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM, (2007) Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med 175: 160-166. Hager DN, Krishnan JA, Hayden DL, Brower RG, (2005) Tidal volume reduction in patients with acute lung injury when plateau pressures are not high. Am J Respir Crit Care Med 172: 1241-1245. Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ, (2012) Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ 344: e2124. Feihl F, Eckert P, Brimioulle S, Jacobs O, Schaller MD, Melot C, Naeije R, (2000) Permissive hypercapnia impairs pulmonary gas exchange in the acute respiratory distress syndrome. Am J Respir Crit Care Med 162: 209-215.
- [Derived] Combes A, Fanelli V, Pham T, Ranieri VM; European Society of Intensive Care Medicine Trials Group and the "Strategy of Ultra-Protective lung ventilation with Extracorporeal CO2 Removal for New-Onset moderate to severe ARDS" (SUPERNOVA) investigators. Feasibility and safety of extracorporeal CO2 removal to enhance protective ventilation in acute respiratory distress syndrome: the SUPERNOVA study. Intensive Care Med. 2019 May;45(5):592-600. doi: 10.1007/s00134-019-05567-4. Epub 2019 Feb 21. PMID 30790030